CLINICAL TRIAL: NCT00673062
Title: Study of the Decongestant Effect of SCH 900538 Compared With Placebo and Pseudoephedrine as Active Control in Subjects With Seasonal Allergic Rhinitis (SAR) Exposed to Pollen in an Environmental Exposure Unit
Brief Title: Study of the Effect of SCH 900538 on Congestion in Subjects With Seasonal Allergic Rhinitis (Study P05031)(COMPLETED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P05031
Record Dates: First submitted 2008-05-05; First posted 2008-05-07 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — Pseudoephedrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- SCH 900538 (Experimental)
  Interventions: Drug: SCH 900538
- Encapsulated pseudoephedrine (Active Comparator): Encapsulated pseudoephedrine (2X30 mg immediate release tablets)
  Interventions: Drug: Pseudoephedrine
- Placebo Capsules (Placebo Comparator)
  Interventions: Drug: Placebo Capsules

INTERVENTIONS:
Drug: SCH 900538 — (4X50mg Capsules)
  Arms: SCH 900538
Drug: Pseudoephedrine — Encapsulated pseudoephedrine (2X30 mg immediate release tablets)
  Other Names: Sudafed
  Arms: Encapsulated pseudoephedrine
Drug: Placebo Capsules — Placebo
  Arms: Placebo Capsules

SUMMARY:
This study is to evaluate the effectiveness of a new drug on congestion in subjects with seasonal allergic rhinitis. This effect will be compared to placebo and to the decongestant, pseudoephedrine.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18 to 65 years of age, of either sex, and of any race.
* Subjects must have a history of SAR due to ragweed for the last two consecutive ragweed seasons.
* Subjects must be skin-test positive for the ragweed pollen allergen used in the Environmental Exposure Unit (pollen chamber at the Screening Visit or within 12 months prior to the Screening Visit.
* Subjects must develop a pre-defined severity of allergy symptoms within 90-minute after entering the pollen chamber during the pollen challenge at the Priming visit (Visit 2), and prior to dosing (Visit 3), in order to qualify for the study.
* Female subjects of childbearing potential must have a negative serum pregnancy test at Screening and a negative urine pregnancy test prior to randomization at the Treatment Visit. Female subjects and female partners of male subjects must be using an acceptable form of birth control during the study.
* Blood pressure and pulse rate must be within normal ranges.

Exclusion Criteria:

* Subjects who have had an upper or lower respiratory tract infection within approximately 28 days (4 weeks) before Priming (Visit 2) and thereafter.
* Subjects who have a dependence upon nasal, oral, or ocular decongestants, nasal topical antihistamines, or nasal steroids, in the opinion of the investigator.
* Subjects with any clinically significant condition or situation, other than the condition being studied that, in the opinion of the investigator, would interfere with the study evaluations or optimal participation in the study.
* Subjects who have used any investigational drugs, including placebo, within 30 days of Screening or for the duration of this stud, or who are participating in any other clinical study.
* Subjects with a history of rhinitis medicamentosa.
* Subjects with a history of anaphylaxis or severe or serious reaction to skin testing.
* Subjects who are being medically treated for any of the following conditions: narrow-angle glaucoma, increased intraocular pressure, urinary retention, hypertension, severe coronary artery disease, ischemic heart disease, diabetes mellitus, hyperthyroidism, renal impairment, or prostatic hypertrophy; current treatment with monoamine oxidase (MAO) inhibitors.
* Subjects with a history of a positive test, or are symptomatic, for HIV, TB (not due to vaccination), and hepatitis B (not due to vaccination) or hepatitis C.
* Subjects with asthma that requires medication other than occasional (<=3 uses per week) use of an inhaled short-acting b-2 agonist.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2008-05; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Average change from baseline in nasal congestion scores over the first 4-hour observation period. | Over the first 4-hour observation period.

SECONDARY OUTCOMES:
Average change from baseline in nasal congestion at each evaluation time point. | Over 12 hours.
Average change from baseline in total symptoms, total symptoms minus congestion, total nasal symptoms, total nasal symptoms minus congestion, total non-nasal symptoms, and individual symptoms scores. | Over the first 4 hour and 12-hour study periods.
Onset of action: defined as the first time point at which a sustained, statistically significant (P<=0.05) reduction relative to placebo in an efficacy variable (eg, nasal congestion) up to a pre-specified time point. | Over the first 4-hours and 12-hour study periods.
Average change from baseline in PNIF over the first 4-hour and 12-hour study periods and at each time point. | Over the first 4-hour and 12-hour study periods.